CLINICAL TRIAL: NCT01650532
Title: The Effects of an 8-Week Yoga Intervention on Cognition and Functional Fitness in Older Adults
Brief Title: Stretching and Yoga Exercise Study
Acronym: SAYExercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Edward McAuley, Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UIUC_IRB_12362
Record Dates: First submitted 2012-07-12; First posted 2012-07-26 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yoga Condition (Experimental): Participants will be instructed to learn yoga postures as well as yoga based breathing and meditative practices by certified yoga instructors. Primary Hatha yoga postures will be performed using props like yoga mats, blocks, belts and blankets. Classes will be held 3 times a week for 8 weeks.
  Interventions: Behavioral: Yoga Condition
- Stretching Condition (Active Comparator): Exercises focusing on stretching and strengthening for all muscle groups will be performed at one-hour long sessions held 3 times a week for 8 weeks. Classes are led by trained exercise specialists.
  Interventions: Behavioral: Stretching Condition

INTERVENTIONS:
Behavioral: Yoga Condition — Classes lasting one hour, held 3 times per week for 8 weeks.
  Arms: Yoga Condition
Behavioral: Stretching Condition — Classes lasting one hour, held 3 times per week for 8 weeks.
  Arms: Stretching Condition

SUMMARY:
The investigators propose to test the effects of an 8-week supervised, site-based, group yoga intervention on cognition and functional fitness in older adults. The SAY Exercise study will compare the yoga group to a stretching group to determine if the program improves attention and cognition, reduces functional limitations, enhances functional performance in everyday activities, as well as psychological health in sedentary older adults between 55-80 years of age. The investigators also propose to assess heart rate variability using a 3-lead EKG and salivary cortisol levels to understand the moderators of the yoga-cognition relationship.

ELIGIBILITY:
Inclusion Criteria:

* 55-80 yrs of age
* Low active: zero to two days of physical activity (>30 minutes per day) per week, in previous six months
* Personal physicians consent to participate in testing and exercise intervention
* Not involved in any other physical activity/exercise research study or cognitive training study.
* Adequate responses to the Telephone interview of Cognitive Status (TICS-M) questionnaire
* Corrected (near and far) acuity of 20/40 or better in both eyes
* Initial depression score on GDS-15 below clinical levels (>5)
* Able to get up and down from the floor
* Comfortable with reading, writing and speaking English

Exclusion Criteria:

* Below 55 or over 80 years of age
* High physical activity levels (more than 2 times per week, >30 minutes, in the last 6 months)
* Regular yoga practitioners (previously or currently practicing for more than 6 months)
* Involved in other physical activity/exercise research study or cognitive training study
* Non-consent of the physician
* Inadequate response on the GDS-15 and TICS-M
* Uncorrected (near and far) acuity of greater than 20/40 in either eye
* Inability to communicate effectively in English
* Intent to be away from the area for a long period of time resulting in more than 2 absences at the exercise sessions

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2012-05; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Changes in cognition as assessed by a neuropsychological battery of computer based and paper pencil tests from baseline to 8 weeks | Baseline - 8 week
  Participants will complete a neuropsychological battery of tasks assessing memory, attention, decision making at baseline (before beginning the program) and at week 8 (after completing the exercise program).

SECONDARY OUTCOMES:
Change in functional fitness from baseline to 8 weeks | Baseline - 8 week
  Participants will complete a battery of physical function tests assessing balance, flexibility, strength and mobility at baseline and week 8.
Change in psychosocial outcomes from baseline to 8 weeks | Baseline - 8 week
  Participants will complete a packet of questionnaires assessing self-esteem, postitive and negative affect including anxiety and depression, self-efficacy and other psychosocial outcomes.
Change in salivary cortisol from baseline to 8 weeks | Baseline - week 8
  Participants will be providing a small saliva sample via a passive drool into a vial. The compound of interest is cortisol (an indicator of body stress).
Change in heart rate variability from baseline to 8-weeks | Baseline - 8 week
  The EKG for each participant will also be recorded in response to a 5 minute unpaced (normal) breathing and 5-minute paced (set to a metronome) breathing. All participants will complete these assessments at baseline and week 8.

CONTACTS AND LOCATIONS:
Overall Officials: Edward McAuley, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Urbana Champaign, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gothe NP, Keswani RK, McAuley E. Yoga practice improves executive function by attenuating stress levels. Biol Psychol. 2016 Dec;121(Pt A):109-116. doi: 10.1016/j.biopsycho.2016.10.010. Epub 2016 Oct 26. PMID 27794449
- [Derived] Gothe NP, McAuley E. Yoga Is as Good as Stretching-Strengthening Exercises in Improving Functional Fitness Outcomes: Results From a Randomized Controlled Trial. J Gerontol A Biol Sci Med Sci. 2016 Mar;71(3):406-11. doi: 10.1093/gerona/glv127. Epub 2015 Aug 22. PMID 26297940